CLINICAL TRIAL: NCT03439475
Title: AMG 714 Expanded Access Program
Status: No longer available | Type: Expanded Access
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: AMG714 Expanded Access Program
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-03

CONDITIONS: Celiac Disease
Keywords: Refractory Celiac Disease Type II
MeSH Terms: conditions — Celiac Disease | interventions — AMG-714

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Biological: AMG 714

SUMMARY:
Expanded access requests for AMG 714 may be considered for adult patients with biopsy proven Refractory Celiac Disease Type II who have failed all available treatment options and do not have EATL. To request access, use Responsible Party contact information provided in this record.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Min Age: 18 Years
Age Groups: Adult, Older Adult